CLINICAL TRIAL: NCT02086929
Title: A Randomized, Double-blind Study Comparing the Efficacy and Safety of Trazodone OAD and Venlafaxine XR in the Treatment of Patients With Major Depressive Disorder.
Brief Title: Trazodone Once a Day in Major Depression Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Aziende Chimiche Riunite Angelini Francesco S.p.A (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 039(C)SC11063
Record Dates: First submitted 2014-03-12; First posted 2014-03-13 (Estimated); Last update posted 2015-12-30 (Estimated); Status verified 2015-12

CONDITIONS: Major Depressive Disorder
Keywords: Trazodone; Venlafaxine; Major depressive disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Trazodone; Venlafaxine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Trazodone (Experimental): 300 mg/day for 8 weeks (including 1 week 150 mg/day of dose-titration). After 3 and 5 weeks of treatment, non responders will have dose increases (in increments of 75 mg/day) till to reach the maximum of 450 mg/day.
  Dosage form: capsule.
  Interventions: Drug: Trazodone
- Venlafaxine XR (Active Comparator): 75 mg/die for 8 weeks. After 3 and 5 weeks of treatment, non responders will have dose increases (in increments of 75 mg/day) till to reach the maximum of 225 mg/day.
  Dosage form: capsule.
  Interventions: Drug: Venlafaxine

INTERVENTIONS:
Drug: Trazodone
  Arms: Trazodone
Drug: Venlafaxine
  Arms: Venlafaxine XR

SUMMARY:
The study objective is to evaluate the efficacy and safety of trazodone OAD vs venlafaxine extended release (venlafaxine XR) after an 8-week treatment period in patients with major depressive disorder.

DETAILED DESCRIPTION:
This randomized, venlafaxine-controlled, double-blind, parallel design study consists of a Pre-Treatment Phase (screening, wash-out) and a double-blind Treatment Phase (randomization to trazodone OAD or to venlafaxine XR, treatment for 8 weeks and tapering for 1 to 3 weeks). During the Pre-Treatment Phase, patients who sign an informed consent form will undergo initial screening. Potential candidates will be instructed to discontinue antidepressants or prohibited medications (wash-out) for a period specific to taper schedule (based on 5 elimination half-lives of the used medication). On the last day of the Pre-Treatment Phase, patients will be evaluated for the final eligibility, and those qualified will be randomly allocated in a 1:1 proportion to trazodone OAD 300 mg/day (1 week of tapering with trazodone OAD 150 mg/day) or to venlafaxine XR 75 mg/day once daily. After 3 and 5 weeks of treatment, subjects will be evaluated for the response. For non responding patients dose increases (in increments of 75 mg/day) will be done till to reach the maximum of 225 mg/day for venlafaxine XR and 450 mg/day for trazodone OAD. Patients non responding to treatment at the final visit will have their study medication tapered from 1 to 3 weeks, according to the maximum dose reached during the study. In order to prevent relapse of depression symptoms, responders at the final visit may continue the treatment. In this case, an unblinded third party Dispenser will open the treatment code and will prescribe the same medication taken by the patients during the trial, according to the formulation available on the market.

ELIGIBILITY:
Inclusion Criteria:

* men and women 18-75 years of age (limits included) with no limitation of race;
* outpatients;
* major depressive disorder according to DSM-IV criteria as assessed using the MINI International Neuropsychiatric Interview;
* 17-item HAMD score > 18 at both screening and baseline visits with a decrease not exceeding 20% between screening and baseline;
* symptoms of depression for at least one month before study entry (screening visit);
* legally capable to give their consent to participate the study, and available to sign and date the written informed consent prior to the inclusion in the study;
* women of childbearing potential must agree not to start a pregnancy from the signature of the informed consent up to 30 days after the last administration of the investigational product.

Exclusion Criteria:

* participation in another trial involving any investigational drug during the past 60 days;
* known hypersensitivity to venlafaxine or trazodone or their excipients;
* use of venlafaxine or trazodone within the previous six months;
* acute, or chronic, or recurrent medical conditions that might affect/jeopardize the study results;
* significant liver disease, defined as active hepatitis or elevated liver enzymes > 3 times the upper boundary of the normal range;
* significant renal disease, defined as urea and/or creatinine > 3 times the upper boundary of the normal range
* myocardial infarction within 6 months prior to start of the double blind treatment;
* positive present history of glaucoma;
* history of risk factors for Torsade de Pointes, such as heart failure, cardiac arrhythmias, bradycardia, cardiac conduction abnormalities, family history of long QT syndrome, cardiac hypertrophy, cardiomyopathy, chronic cardiac insufficiency;
* values of electrolytes (sodium, potassium, calcium, magnesium, chloride) outside the normal laboratory range and judged clinically relevant by the Investigator;
* concomitant treatment with drugs known for QT prolongation, or with drugs producing hypokalemia, or diuretics;
* QTcF values higher than 450 msec in the ECG performed at the screening;
* history of major depression resistant to medical treatments (previous failure to respond to two consecutive antidepressants of different classes used for a sufficient length of time at appropriate doses);
* history of seizure events other than a single childhood febrile seizure;
* history of alcohol or psychoactive substance abuse or addiction (except caffeine or nicotine) during the last year as defined by DSM-IV criteria;
* positive urine drug screen for CNS-active drugs (cocaine, opioids, amphetamines and cannabinoids) at Visit 1 (screening);
* acute risk of suicide (HAMD, criterion 3 with a value > 3);
* presence of any primary psychiatric disorder other than major depression;
* history or presence of bipolar disorder, any psychotic disorder, mental disorder due to general medical conditions;
* pregnancy, lactation, or female with a positive urine pregnancy test result at Visit 1 (Screening);
* electroconvulsive therapy (ECT) within 30 days prior to the screening visit;
* use of antipsychotic drugs within two months prior to the baseline visit (Visit 2);
* use of any anxiolytic or sedative hypnotic drug within seven days prior to the baseline (Visit 2) and during the study. Exception is stable low doses of benzodiazepines for insomnia (if taken by the patient more than two weeks before the Treatment Phase);
* use of any psychotropic drug or substance with central nervous system effects within seven days prior to the baseline visit (Visit 2);
* use of any non-psychotropic drug with psychotropic effects (e.g. alpha-adrenergic blockers) within seven days prior to the baseline visit (visit 2), unless a stable dose of the drug has been maintained for at least one month (three months for thyroid or hormonal medications) before the baseline visit (visit 2);
* concomitant treatment with CYP3A4 inhibitors (e.g. ketoconazole, ritonavir, indinavir);
* hyperthyroidism, even if pharmacologically corrected;
* start or discontinuation of psychotherapy within 6 weeks prior to screening;
* clinically significant abnormalities on physical examination, vital signs, ECG, laboratory tests at the screening visit;
* high blood pressure (supine systolic blood pressure > 160 mmHg or supine diastolic blood pressure > 90 mmHg) at screening or baseline, either untreated or under treatment with antihypertensives
* inability to comply with the protocol requirements, instructions and study-related restrictions; e.g. uncooperative attitude, inability to return for study-visits, and improbability of completing the clinical study;
* vulnerable subjects (e.g. persons kept in detention);
* if subject is the Investigator or his/her deputies, first grade relative, research assistant, pharmacist, study coordinator, other staff of relative thereof directly involved in the conduct of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 364 (Actual)
Dates: Start 2012-12; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Hamilton Depression Rating Scale (HAMD) score | Day 56
  Mean change from baseline (Day 0) in HAMD score at Day 56.

SECONDARY OUTCOMES:
Montgomery-Asberg Depression Rating Scale (MADRS) score | Day 56
  Mean change from baseline (Day 0) in MADRS score at Day 56.
Clinical Global Impression (CGI) Severity of Illness score | Day 56
  CGI-Severity of Illness improvement at Day 56.
Clinical Global Impression (CGI) Global improvement score | Day 56
  CGI-Global improvement at Day 56.
Percentage of responders | Day 56
  Rate of patients with a 50% decrease with respect to baseline on the HAMD score at Day 56.
Percentage of patients with remission | Day 56
  Rate of patients with a HAMD score <or= at Day 56.
Safety profile of trazodone OAD compared to venlafaxine XR | 11 weeks
  Safety and tolerability will be assessed through adverse events monitoring, physical examinations and monitoring of vital signs, body weight, clinical laboratory tests, ECG.

CONTACTS AND LOCATIONS:
Overall Officials: Filippo Bogetto, MD, Principal Investigator — Department of Neuroscience University of Turin - Italy
Locations (32):
- Austria (2):
  - Institute für Psychosomatik, Vienna
  - AKH Wien, Vienna
- Czechia (10):
  - PRAGTIS, s.r.o., Prague, Prague
  - Psychiatry Trial, s.r.o., Prague, Prague
  - MEDICAL SERVICES PRAGUE, s.r.o., Prague, Prague
  - Neuropsychiatrie s.r.o., Prague, Prague
  - Saint Anne, s.r.o., Brno-mesto
  - SUPERVIZE, s.r.o., Kutná Hora
  - BIALBI s.r.o., Litoměřice
  - Fakultni Nemocnice Olomouc, Klinika Psychiatrie, Olomouc
  - MUDr. Eva Soukupová-Psychiatrická praxe, s.r.o., Pilsen
  - NZZ- MUDr. Jaroslav Hronek, psychiatrická ambulance, Pilsen
- Italy (6):
  - UOPI di Psichiatria Azienda Ospedaliero Universitaria Policlinico Vittorio Emanuele, Presidio "Gaspare Rodolico", Catania, Catania
  - Clinica Psichiatrica Nuovo Ospedale S. Salvatore Università degli Studi del L'Aquila, L’Aquila, L'Aquila
  - Ospedale Santa Maria della Misericordia Unità di Degenza Psichiatrica-SPDC, Perugia, Perugia
  - Azienda Ospedaliera Sant'Andrea Università La Sapienza Unità Operativa Complessa di Psichiatria, Rome, Rome
  - AOUS-Azienda Ospedaliera Universitaria Senese Policlinico Santa Maria alle Scotte Clinica Psichiatrica Universitaria, Siena, Siena
  - Department of Neurosciences University of Turin, Turin, Turin
- Romania (7):
  - Quantum Medical Center Srl, Bucharest
  - Spitalul clinic de psihiatrie "Prof. Dr. Al. Obregia"/Sectia 13, Bucharest
  - Spitalul Clinic de Psihiatrie "Prof. Dr. Al. Obregia"/Sectia 1, Bucharest
  - Spitalul Clinc de Urgenta Militar "Dr. Stefan Odobleja", Craiova, Craiova
  - Spital Clinic de Psihiatrie SOCOLA / Iasi, Iași
  - Spitalul de Psihiatrie "Dr. Gh.Preda" Sibiu, Sibiu
  - Spitalul Clinc Judetean Mures, Centrul de Sanatate Mintala, Târgu Mureş
- Slovakia (6):
  - Psychiatricka ambulancia, Bratislava
  - MENTUM, s.r.o., Bratislava
  - EPAMED, s.r.o., Košice
  - Psychiatricka nemocnica, Michalovce
  - Psycholine, s.r.o., Rimavská Sobota
  - Psychiatricke oddelenie, NsP sv Barbory Roznava, Rožňava
- Instituto de Investigacion y Asistencia Psiquiatrica - IIAP, Madrid, Spain

REFERENCES:
- See also: Sponsor's website — http://www.angelinipharma.com